CLINICAL TRIAL: NCT04890912
Title: Stereotactic Pelvic Adjuvant Radiation Therapy in Cancers of the Uterus II: A Phase II Randomized Controlled Trial
Brief Title: Stereotactic Pelvic Adjuvant Radiation Therapy in Cancers of the Uterus II
Acronym: SPARTACUSII
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Royal Victoria Hospital, Canada (Other); Credit Valley Hospital (Other); London Regional Cancer Program, Canada (Other)
Responsible Party: Principal Investigator, Dr. Eric Leung, Principal Investigator, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPARTACUS II
Record Dates: First submitted 2021-05-05; First posted 2021-05-18 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Endometrial Cancer
Keywords: endometrial cancer; uterine cancer
MeSH Terms: conditions — Endometrial Neoplasms; Uterine Neoplasms | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Fractionation Pelvic Radiation (Active Comparator): Patients randomized to the conventional fractionation arm will be treated with intensity-modulated or volumetric arc therapy technique as per standard protocol.
  Interventions: Radiation: Conventional Fractionation
- Stereotactic Hypofractionated Radiation (Experimental): Patients randomized to hypofractionation will be treated the stereotactic hypofractionated technique.
  Interventions: Radiation: Hypofractionation

INTERVENTIONS:
Radiation: Conventional Fractionation — Dose prescribed is 45 Gy in 25 fractions (1.8 Gy per fraction) delivered daily over 5 weeks.
  Arms: Conventional Fractionation Pelvic Radiation
Radiation: Hypofractionation — Dose prescribed is 30 Gy in 5 fractions (6 Gy per fraction) delivered every other day over 11 days. There will be a minimum of 36 hours and maximum of 96 hours between fractions. The entire course of treatment should be completed within no less than 10 days.
  Arms: Stereotactic Hypofractionated Radiation

SUMMARY:
Adjuvant radiotherapy (RT) plays an important role in reducing the risks of local recurrence after surgery in uterine cancers. Standard adjuvant pelvic radiation treatment targets the pelvic lymph nodes, the post-operative bed, and the upper vagina and is typically treated with intensity modulated radiation therapy (IMRT) which has been shown to improve patient reported gastrointestinal (GI) and genitourinary (GU) toxicities. Although pelvic radiation has been shown to be effective at decreasing locoregional recurrences, patient quality of life and experience can be significantly impacted as pelvic RT comprises of daily radiation for 25 daily treatments, which can be a substantial burden on patients with this disease. Hypofractionated radiotherapy to a dose of 30 Gy in 5 fractions (6 Gy given every other day) for adjuvant radiation treatment in uterine cancer is hypothesized to result in similar rates of acute gastrointestinal toxicities as conventional fractionated radiation.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with histologically confirmed endometrial adenocarcinoma, serous or clear cell carcinoma.
2. Patient is a candidate for adjuvant pelvic radiation for uterine cancer (+/- vault brachytherapy), meeting one of the following conditions:

   High grade histology (including serous and clear cell) OR Outer-half myometrial invasion and International Federation of Gynecology and Obstetrics (FIGO) grade 1-2 OR FIGO stage II - III.
3. Patients who are to receive adjuvant systemic therapy sequentially in addition to pelvic radiotherapy will be eligible.
4. Age ≥18 years.
5. Patient is willing and able to give informed consent to participate in this clinical trial.

Exclusion Criteria:

1. Patient has had prior pelvic radiotherapy.
2. Patient has a contraindication to pelvic radiotherapy, such as but not limited to a connective tissue disease or inflammatory bowel disease.
3. Patient planned for concurrent chemoradiation therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Acute bowel toxicity | Baseline to 2 years following RT completion
  To compare the acute bowel toxicities associated with hypofractionated vs conventional adjuvant pelvic radiation as measured by the The Expanded Prostate Cancer Index Composite (EPIC) questionnaire.

SECONDARY OUTCOMES:
Acute bowel toxicities | Baseline to 2 years following RT completion
  To compare the acute bowel toxicities associated with hypofractionated treatment and conventional fractionation in adjuvant pelvic radiation for endometrial cancers using the Common Terminology Criteria for Adverse Events (CTCAE v5.0) criteria.
Acute urinary toxicities through CTCAE | Baseline to 2 years following RT completion
  To compare the acute urinary toxicities associated with hypofractionated treatment and conventional fractionation in adjuvant pelvic radiation for endometrial cancers using the Common Terminology Criteria for Adverse Events (CTCAE v5.0) criteria.
Acute urinary toxicities through EPIC | Baseline to 2 years following RT completion
  To compare the acute urinary toxicities associated with hypofractionated treatment and conventional fractionation in adjuvant pelvic radiation for uterine cancer as measured by EPIC.
Local- regional failure | Baseline to 2 years following RT completion
  To compare presence of tumour through physical exam or radiologic imaging between hypofractionated treatment and conventional fractionation.
Disease-free survival | Baseline to 2 years following RT completion
  To compare disease-free survival of hypofractionated treatment and conventional fractionation
Quality of life using EORTC QLQ-30 and endometrial module (EN-24) | Baseline to 2 years following RT completion
  To compare the effect of hypofractionated treatment and conventional fractionation on quality of life using the using EORTC (European Organisation for Research and Treatment of Cancer) core questionnaire (QLQ-C30) with EN-24 companion.
Correlation of GU toxicity, EORTC, and EPIC | Baseline to 2 years following RT completion
  To measure correlations between GU toxicity and EORTC questionnaire versus GU toxicity and EPIC questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Leung, MD, Principal Investigator — Sunnybrook Health Sciences Centre; Kathy Han, MD, Principal Investigator — Princess Margaret Cancer Centre; Adam Gladwish, MD, Principal Investigator — Royal Victoria Hospital, Belfast
Locations (5):
- Canada (5):
  - Royal Victoria Hospital, Barrie, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No